CLINICAL TRIAL: NCT01063452
Title: Impact of Atkinson Product Design Urinary Slide Valve Versus Standard Catheter Drainage System on Social Functioning
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This trial was never initiated due to inability to obtain the device
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Dr. Manoj Monga, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Truvalve
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Urinary Catheterization; Urinary Tract Infections
Keywords: Urinary Catheterization; Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Truvalve (Experimental): Atkinson Product Design urinary slide valve on the catheter
  Interventions: Device: Truvalve
- Control (Active Comparator): Drainage bag on the catheter
  Interventions: Other: Control (catheter drainage bag)

INTERVENTIONS:
Device: Truvalve — Atkinson Product Design urinary slide valve
  Arms: Truvalve
Other: Control (catheter drainage bag) — urinary catheter drainage bag
  Arms: Control

SUMMARY:
The primary objective of this study is to evaluate the impact of the Atkinson Product Design urinary slide valve on patient morbidity and freedom as measured by impact on activities of daily living (ADL) and quality of life (QOL). Secondary objectives include assessing the impact of the device on bacteruria and evaluating the impact of the primary treatment on ADL and QOL.

DETAILED DESCRIPTION:
Several indications exist in urologic practice where urinary drainage via a urethral catheter is required and an estimated 4 million patients in the United States undergo urinary catheterization per year.(1) Though it is common for urine to be continually collected in a bag attached to the catheter by plastic tubing, catheter valves offer an alternative method of storing and voiding urine. Catheter valves are small devices that fit into the external end of the urethral catheter. Rather than continuous drainage, urine is stored in the bladder and emptied on regular intervals by opening the valve.

This method of drainage may offer several benefits including preserving bladder capacity, function and tone, reducing catheter blockage in cases of urine bacterial colonization, and decreasing traction forces on the bladder neck by removing the downward weight of a collecting bag.(2-4) The use of a catheter valve may offer improvements in social functioning and mobility.(5) Studies to date suggest that catheter valves are well tolerated by patients, but these studies have used non-standardized questionnaires and have not assessed overall quality of life.(5, 6) Additionally, there may be an associated cost benefit to utilizing catheter valves compared to drainage bags.(5)

Further study in this area, focusing on quality of life and social functioning, will enable the clinician to better counsel patients on the risks and benefits of the various methods of urinary drainage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing brachytherapy or cryotherapy for prostate cancer
2. Patients undergoing thermal therapy for benign prostatic hyperplasia
3. Patients undergoing catheterization to relieve urinary retention

Exclusion Criteria:

1. Patients with neurogenic bladder
2. Patients with urinary tract infection
3. Patients with gross hematuria
4. Patients undergoing surgery with risk of urinary leak (ex: urethroplasty, radical prostatectomy, bladder repair)
5. Female patients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the impact of the Atkinson Product Design urinary slide valve on patient morbidity and freedom as measured by impact on activities of daily living (ADL) and quality of life (QOL). | 1 month after catheter removal

SECONDARY OUTCOMES:
Secondary objectives include assessing the impact of the device on bacteruria and evaluating the impact of the primary treatment on ADL and QOL. | At time of catheter removal

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Monga, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Urology Associates, Edina, Minnesota
  - University of Minnesota, Minneapolis, Minnesota